CLINICAL TRIAL: NCT04293653
Title: Protocol for Patients Above 75 Years Undergoing Emergency Laparotomy
Acronym: (ProPEL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REK7110
Record Dates: First submitted 2020-01-02; First posted 2020-03-03 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-08

CONDITIONS: Frailty; Surgery--Complications; Outcome, Fatal; Frail Elderly Syndrome; Post-Op Complication; Gastro-Intestinal Disorder
MeSH Terms: conditions — Frailty; Postoperative Complications; Digestive System Diseases | interventions — Clinical Protocols; Laparoscopy

STUDY DESIGN:
Intervention Model Description: A care-bundle developed for patients above 75 years undergoing emergency abdominal surgery will be investigated, and the results will be compared to a group of historical controls operated at Haukeland University Hospital in 2016-2017, using 30-day mortality as the primary outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Care bundle (Experimental): Patients above 75 years where emergency surgery is indicated, deemed fit for surgery, will be included in a perioperative care-bundle. While waiting for surgery, patients will be monitored and optimized if their condition deteriorates. Antibiotics will be administered if indicated. Surgery will be delivered within 2h to 72h, depending on the suspected abdominal pathology and the patient's clinical condition.
  Interventions: Other: Protocol for patients above 75 undergoing emergency laparotomy or laparoscopy

INTERVENTIONS:
Other: Protocol for patients above 75 undergoing emergency laparotomy or laparoscopy — See above section

SUMMARY:
In the ProPEL study the effect of a protocol designed for elderly patients about to undergo emergency abdominal surgery will be investigated. The protocol addresses issues of both frailty and ceiling-of -care decisions.

DETAILED DESCRIPTION:
In the "ProPEL" study, investigators will test the effect of a care bundle designed for patients aged ≥75 years undergoing emergency laparotomy/laparoscopy. An interdisciplinary team of anesthetists, intensivists, surgeons, and geriatricians developed the care bundle, and the essential elements are frailty scoring, surveillance and optimization of patients, surgical treatment within predefined criteria, and postoperative delirium monitoring.

Preoperatively, patients with abdominal pathology requiring emergency surgery will be evaluated for frailty by the surgical team, using standardized frailty scores. Palliative care could be an alternative to surgery in very frail patients. The decision to not perform surgery is a clinical decision made with the patient and/or relatives in a shared decision-making process. Frailty scoring can assist in this procedure.

The effect of the care-bundle will be compared to a historical cohort, using 30-day mortality as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

- Patients above 75 years with clinical suspicion of abdominal condition requiring surgery

Exclusion Criteria:

* Former inclusion in "ProPEL"
* Surgery for incarcerated hernia without laparotomy
* Appendectomy without laparotomy
* Palliative surgery for already known inoperable gastrointestinal tumor
* Palliation without surgical treatment
* Vascular surgery

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Composite score of 30-day mortality and postoperative complications | Up to 30 days after the performance of emergency abdominal surgery
  Composite score will be calculated using the Comprehensive Complication Index ranging from 0 points (uneventful postoperative recovery) to 100 points (postoperative death). One investigator will review the patient's medical record postoperatively to investigate if any medical complication has occurred. Complications are defined according to the EPCO definitions and graded according to the Clavien-Dindo classification system.

SECONDARY OUTCOMES:
Postoperative complications | up to 90 days after date of emergency surgery
  Number of patients having a postoperative complication as defined by the European Perioperative Clinical Outcome Definitions (EPCO) will be reported. The EPCO definitions state universal description of various common postoperative complications, like f.ex pulmonary complications, major adverse cardiac events, urinary tract infections and so on. Thus, postoperative complications are reported in a uniform way.
  We will grade complications according to the Clavien-Dindo classification. According to this classification postoperative complications are graded from 1 to 5, where 1 indicates least severity of complication and 5 indicating worst severity. We will report number of patients having complications from grade 2 to grade 5.
Frequency of post-operative delirium | up to 30 days after emergency surgery
  Number of patients having postoperative delirium as defined by the screening tool 4 AT. On this 4-item screening tool for delirium patients are scored from 0 (minimum) up to 12 points (maximum). Screening for delirium is positive if score is 4 or above.
Length of stay in hospital after EAS | up to 90 days after emergency surgery
  Number of days spent in hospital after EAS
Patients' Level of independency as measured by the Barthel Activity of Daily Living Index before surgery and one year after surgery | Patients will be assessed with the BArthel ADL-index when admitted to hospital and again one year after emergency abdominal surgery.
  Activity of Daily Living (ADL) is measured using the Barthel ADL-index (Norwegian Version), a validated 10-item questionnaire. In this scale the patients level of functioning is described and assigned from 0 to 20 points. Zero points indicate total dependency and 20 points indicate Complete independency in Activities of Daily Living.
Level of care at discharge from hospital and one year after EAS | 1 year after EAS.
  Number of patients discharged to own home after EAS. Number of patients discharged to nursing home after EAS. Number of patients living in own home or in nursing home one year after EAS.
1-year mortality | From time of EAS performed and up to 1 year
  Number of deaths within 1 year after emergency abdominal surgery (EAS)
Days at home in first postoperative year | From date of discharge from hospital after EAS and up to one year postoperatively
  Number of days living in own home first year after EAS
Readmissions after EAS | From 8 hours after primary discharge from hospital after EAS until 30 days after primary discharge.
  Number of patients readmitted to hospital after first being discharged from hospital after EAS
Patient Reported Outcome Measures (PROM)one year after EAS | One year after procedure performed (EAS).
  Patients report on own Health performance as measured by the 36-Item Short Form Survey. In this survey patients subjective health status is described using 36 standardized questions. Patients will also be asked about their willingness to undergo same procedure again, if indicated.
5-year survival | From inclusion in study and up to five years after EAS.
  Number of Deaths occurring within 5 years after EAS
30-day mortality in all patients with indication to undergo surgery | Time (days) up to 30 days after treatment decision (palliation or surgery) is made
  30-day mortality rate in palliative and operated patients

OTHER OUTCOMES:
3-year survival | Time (days) from end of index surgery and up to 3 years after EAS.
  Number of deaths occuring within 3 years after EAS

CONTACTS AND LOCATIONS:
Overall Officials: Ib Jammer, MD, PhD, Principal Investigator
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No